CLINICAL TRIAL: NCT06079866
Title: Assessment of the Seal, Comfort, Usability, and Performance of the Oran Park Mask System in the Home Environment
Brief Title: Oran Park Mask External Clinical Study (3) Marketing Claims Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SLP-23-04-01; D646-159 (Other: ResMed)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Both masks (Oran Park Mask and Evora Mask (Mask A and Mask B)) will be worn for a period of 7 nights sequentially. Participants will complete a series of questionnaires upon completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Mask A (Oran Park Mask) then Mask B (Evora Mask) (Other): Participants will be randomized as to the order they will trial Mask A and Mask B. This arm will first use the Oran Park mask for 7 days and then use the Evora Mask for 7 days.
  Interventions: Device: Mask A (Oran Park Mask) then Mask B (Evora Mask)
- Mask B (Evora Mask) then Mask A (Oran Park Mask) (Other): Participants will be randomized as to the order they will trial Mask A and Mask B. This arm will first use the Evora mask for 7 days and then use the Oran Park mask for 7 days.
  Interventions: Device: Mask B (Evora Mask) then Mask A (Oran Park Mask)

INTERVENTIONS:
Device: Mask A (Oran Park Mask) then Mask B (Evora Mask) — Mask A (Oran Park Mask) for 7 days followed by Mask B (Evora Mask) for 7 days
  Arms: Mask A (Oran Park Mask) then Mask B (Evora Mask)
Device: Mask B (Evora Mask) then Mask A (Oran Park Mask) — Mask B (Evora Mask) for 7 days followed by Mask A (Oran Park Mask) for 7 days.
  Arms: Mask B (Evora Mask) then Mask A (Oran Park Mask)

SUMMARY:
The goal of this prospective, randomized, open label, cross over study to assess the seal, comfort, usability, and performance of the prototype Oran Park mask system (referred to as Mask A in this study protocol) in the home environment. Comparisons will be made against Fisher & Paykel's Evora Full mask system (referred to as Mask B in this study protocol, an FDA cleared benchmark mask) and the participant's own mask.

Patients diagnosed with Obstructive Sleep Apnea and are current CPAP users on a tube down full-face mask system will be recruited to the study to evaluate the Oran Park mask system and the Evora Full mask system for up to 7 nights each, in the home environment, whilst using their own CPAP device.

The overall purpose is to evaluate the performance of the prototype Oran Park mask system compared to an FDA cleared benchmark mask (Evora Full) in relation to seal, comfort, usability, ease of use, preference, AHI, and objective therapy data.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who can read and comprehend English
* Participants who ≥ 18 years of age
* Participants being treated for OSA for ≥ 12 months
* Participants who have met CMS compliance for CPAP therapy over the last 3 months
* Participants who have been using a ResMed cloud connected AirSense10 or AirSense 11 device compatible with AirView, for more than 12 months
* Participants currently using a suitable mask system*
* Participants who can trial the masks for up to 7 nights each

  * Note*: Suitable mask system includes any tube down full face mask (e.g. AirFit F30, AirFit F20, AirTouch F20, AirFit F10, Quattro Air, Quattro Fx, Mirage Quattro, Simplus, Amara, Amara Gel, Comfort gel Full Face Mask, Evora Full)

Exclusion Criteria:

* Participants using Bi-level flow generators
* Participants who are or may be pregnant
* Participants with a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants who or whose bed partner has implantable metallic implants in the head, neck and chest region affected by magnetic fields (Non-ferrous implants may be acceptable)
* Participants who use a rental unit for AirSense 10 or AirSense 11 device
* Participants believed to be unsuitable for inclusion by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
11 point Likert Scale Questionnaire | 7 days
  • Subjective scores will be collected from subjects on each attribute being assessed (e.g. seal, comfort, ease of use etc.). Scores will be collected using an 11-point Likert Scale Questionnaire. Minimum value will be zero. Maximum value will be 10. A higher score indicates better outcomes. A score of 10 is considered very favorable, and a score of 0 is very unfavorable.

SECONDARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 7 days
  • The AHI recorded by the subject's PAP device while using their own mask will be compared to the AHI recorded by the subject's PAP device while using the Oran Park mask and the Evora Mask. The AHI will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.
Leak | 7 days
  The median air leak (L/minute) recorded by the subject's PAP device while using their own mask will be compared to the median air leak (L/minute) recorded by the subject's PAP device while using the Oran Park mask and the Evora mask. The median air leak will be obtained from the ResMed AirView Compliance Reports downloaded during the study visits.
Pressure Differences | 7 days
  The median air pressure (cmH2O) used during PAP therapy recorded by the subject's PAP device while using their own mask will be compared to the median air pressure (cmH2O) recorded by the subject's PAP device while using the Oran Park mask and the Evora mask. The median air pressure levels will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.
Compliance | 7 days
  The subject's average daily hours of use of PAP therapy recorded by the subject's PAP device while using their own mask will be compared to the average daily hours of use recorded by the subject's PAP device while using the Oran Park mask and the Evora mask. The average daily hours of use will be obtained from the ResMed AirView Compliance Reports downloaded from the subject's PAP device during the study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Uhles, Principal Investigator — Clayton Sleep Institute; Betsy Dauphin, Principal Investigator — Sleep Data
Locations (2):
- United States (2):
  - Sleep Data, San Diego, California
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No